CLINICAL TRIAL: NCT06500572
Title: Ultrasound Guided, Landmark Guided Intercostobrachial Nerve Block Versus Serratus Plane Block After Supraclavicular Plexus Block for Anesthesia in Creation of Arteriovenous Fistula in the Medial Side of the Arm: A Randomized Trial
Brief Title: Landmark Guided Intercostobrachial Nerve Block Versus Serratus Plane Block After Supraclavicular Plexus Block for Anesthesia in Creation of Arteriovenous Fistula in the Medial Side of the Arm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Zakarea Wfa, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264PR77/5/24
Record Dates: First submitted 2024-07-08; First posted 2024-07-15 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Intercostobrachial Nerve Block; Serratus Plane Block; Supraclavicular Plexus Block; Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Landmark Guided Intercostobrachial Nerve Block (Active Comparator): In addition to the supraclavicular plexus block, the intercostobrachial nerve block block will be performed without ultrasound guidance and based on the traditional method using superficial anatomy and nerve pathway by subcutaneous injection of 20 mL of bupivacaine 0.25% at the site of the pulse.
  Interventions: Other: Landmark Guided Intercostobrachial Nerve Block
- Ultrasound Guided Intercostobrachial Nerve Block (Experimental): The patient's head will be turned to the opposite side while the patient is in the supine position and the shoulder to be treated will be elevated 5- 10 cm. The high-frequency linear ultrasound probe (12-4 MHz) and the region to be treated will be prepared in sterile conditions and placed transversely across the external jugular vein at 3-4 cm above the clavicle. Between the anterior and middle scalene muscles, the imaging of the brachial plexus showed three to five hypoechoic circles. The entry will be in-plane technique using an 80-mm block needle from lateral to medial. After confirming the needle insertion site with 2 mL saline solution, a 20 mL bupivacaine 0.25% will be administered.
  Interventions: Other: Ultrasound Guided Intercostobrachial Nerve Block
- Serratus Plane Block (Experimental): The patient will be placed in the lateral decubitus position with the area to be treated on the upper side. The high-frequency linear ultrasound probe and the region to be treated will be sterilized. The ultrasound probe will be placed on the anterior line at the level of fourth and fifth ribs. Images of the muscle's latissimus dorsi and serratus anterior, the ribs, and the pleura will be obtained. Subsequently, with the in-plane technique, an 80-mm block needle will be advanced between the latissimus dorsi and the serratus muscles planes in a caudal to the cranial direction. There is no blood or air in aspiration. After confirming the location of the needle with 2 mL of saline solution, (20 mL of bupivacaine 0.25%) will be administered between the two muscles.
  Interventions: Other: Serratus Plane Block

INTERVENTIONS:
Other: Landmark Guided Intercostobrachial Nerve Block — In addition to the supraclavicular plexus block, the intercostobrachial nerve block block will be performed without ultrasound guidance and based on the traditional method using superficial anatomy and nerve pathway by subcutaneous injection of 20 mL of bupivacaine 0.25% at the site of the pulse.
  Arms: Landmark Guided Intercostobrachial Nerve Block
Other: Ultrasound Guided Intercostobrachial Nerve Block — The patient's head will be turned to the opposite side while the patient is in the supine position and the shoulder to be treated will be elevated 5- 10 cm. The high-frequency linear ultrasound probe (12-4 MHz) and the region to be treated will be prepared in sterile conditions and placed transversely across the external jugular vein at 3-4 cm above the clavicle. Between the anterior and middle scalene muscles, the imaging of the brachial plexus showed three to five hypoechoic circles. The entry will be in-plane technique using an 80-mm block needle from lateral to medial. After confirming the needle insertion site with 2 mL saline solution, a 20 mL bupivacaine 0.25% will be administered.
  Arms: Ultrasound Guided Intercostobrachial Nerve Block
Other: Serratus Plane Block — The patient will be placed in the lateral decubitus position with the area to be treated on the upper side. The high-frequency linear ultrasound probe and the region to be treated will be sterilized. The ultrasound probe will be placed on the anterior line at the level of fourth and fifth ribs. Images of the muscle's latissimus dorsi and serratus anterior, the ribs, and the pleura will be obtained. Subsequently, with the in-plane technique, an 80-mm block needle will be advanced between the latissimus dorsi and the serratus muscles planes in a caudal to the cranial direction. There is no blood or air in aspiration. After confirming the location of the needle with 2 mL of saline solution, (20 mL of bupivacaine 0.25%) will be administered between the two muscles.
  Arms: Serratus Plane Block

SUMMARY:
This study aims to compare the role of ultrasound-guided and landmark-guided intercostobrachial nerve block and serratus plane block after supraclavicular plexus block for anesthesia in the creation of an arteriovenous fistula in the medial side of the arm.

DETAILED DESCRIPTION:
Brachial plexus block (BPB) is usually utilized for proximal arm arteriovenous access creation. It has been suggested that supraclavicular brachial plexus block (SCPB) could be an alternative and provide comparable effective anesthesia and postoperative analgesia for arm surgery, with a reduced incidence of adverse events, including hemidiaphragmatic paresis.

By performing SCPB, the inner part of the arm is not completely anesthetized because this part of the arm is innervated by the lateral cutaneous branch of the second intercostal nerve (intercostobrachial nerve (ICBN)) and the medial branch of the brachial cutaneous nerve.

Serratus plane block (SPB) was first defined in 2013 by Blanco et al. This block provides anesthesia and analgesia in the hemi-thorax, where it is applied to block the thoracic intercostal nerves, in addition to the axillary region and shoulder posteriorly.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Scheduled for creation of arteriovenous fistula in the medial side of the arm.

Exclusion Criteria:

* Allergy to local anesthetics.
* Drug addiction.
* Coagulation abnormalities.
* Body Mass Index (BMI)≥35 kg/m2.
* Upper extremity neuropathy.
* Vasculitis.
* Unstable hemodynamics.
* History of seizures or mental illness.
* Severe heart, kidney, and liver diseases.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-07-13 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Percent of patients who needed local anesthetic supplementation | Intraoperatively
  Number of patients who needed local anesthetic supplementation will be recorded.

SECONDARY OUTCOMES:
Total amount of morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the visual analog scale (VAS) > 3 to be repeated after 30 min if pain persists until the VAS < 4. VAS will be assessed at 0, 2, 4, 8, 12 and 24 h postoperatively.
Patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.